CLINICAL TRIAL: NCT04693416
Title: SMART Trial: Reducing Stigma Towards Opioid Use Disorder on the Intrapersonal and Interpersonal Levels
Brief Title: SMART Trial: Intrapersonal and Interpersonal Stigma Reduction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Karen Derefinko, PhD, Assistant Professor, University of Tennessee
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-07852; 3R61AT010604-01S1 (NIH)
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Results first posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Stigma, Social; Opioid Use; Opioid-use Disorder; Substance Use Disorders
Keywords: opioid use disorder; substance use disorder; stigma
MeSH Terms: conditions — Social Stigma; Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrapersonal Stigma Reduction (Experimental): The intervention will include education about substance use disorders (diagnosis, prognosis, and treatment), goal setting to assist the individual in preparing for change, and decisional balance to assist the individual in measuring the costs and benefits about disclosure of mental health problems and exercises to practice how to disclose. Facilitation of an intake assessment for treatment will be offered (with assistance in making the appointment, getting transportation and childcare, and securing a pro-bono status at a outpatient treatment facility).
  Interventions: Other: Intrapersonal Stigma Reduction
- Interpersonal Stigma Reduction (Experimental): The intervention for family members and support persons of enrolled intrapersonal participants will include education about substance use disorders (diagnosis, prognosis, and treatment), stigma reduction, and how to provide support for someone with substance use disorder.
  Interventions: Other: Interpersonal Stigma Reduction

INTERVENTIONS:
Other: Intrapersonal Stigma Reduction — Brief intervention for stigma reduction
  Arms: Intrapersonal Stigma Reduction
Other: Interpersonal Stigma Reduction — Brief intervention for support persons of intrapersonal intervention participants.
  Arms: Interpersonal Stigma Reduction

SUMMARY:
The goal of this project is to develop a multicomponent stigma reduction intervention to address intrapersonal (individual) stigma regarding Opioid Use Disorder (OUD). The intervention will address this cost/benefit evaluation among individuals known to face intersecting stigma of OUD and African American race, with treatment elements chosen explicitly to increase the value of treatment using salient forms of reward, and to ease perceived costs through explicit services in an effort to encourage the occurrence of the first treatment visit for OUD.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Identify as African American, Black, or mixed race
* Identify as someone with a substance use disorder who is not currently in treatment OR a support person of someone enrolled
* Access to a telephone for follow-up assessment
* Reside in the Memphis, TN area

Exclusion Criteria:

* Unable to understand consent procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen J Derefinko, PhD, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Background] Smith LR, Earnshaw VA, Copenhaver MM, Cunningham CO. Substance use stigma: Reliability and validity of a theory-based scale for substance-using populations. Drug Alcohol Depend. 2016 May 1;162:34-43. doi: 10.1016/j.drugalcdep.2016.02.019. Epub 2016 Feb 26. PMID 26972790
- [Background] Palamar JJ. An examination of beliefs and opinions about drug use in relation to personal stigmatization towards drug users. J Psychoactive Drugs. 2013 Nov-Dec;45(5):367-73. doi: 10.1080/02791072.2013.843044. PMID 24592661
- [Background] Palamar JJ, Kiang MV, Halkitis PN. Development and psychometric evaluation of scales that assess stigma associated with illicit drug users. Subst Use Misuse. 2011;46(12):1457-67. doi: 10.3109/10826084.2011.596606. Epub 2011 Jul 18. PMID 21767076

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in the intrapersonal intervention were recruited from community centers in the target area. Participants in the interpersonal intervention were support persons referred by the participants in the intrapersonal intervention.
Period: Overall Study
Arm/Group | Intrapersonal Stigma Reduction | Interpersonal Stigma Reduction
Started | 50 | 21
Completed | 37 | 21
Not Completed | 13 | 0
Not completed — Lost to Follow-up | 13 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intrapersonal Stigma Reduction | Interpersonal Stigma Reduction | Total
Number analyzed (Participants) | 50 | 21 | 71
Age, Continuous [Mean (Full Range); unit: years] | 42.9 [22 to 66] | 36.3 [19 to 55] | 41.0 [19 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 15 | 40
  Male | 25 | 6 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 50 | 21 | 71
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 50 | 21 | 71
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 21 | 71

OUTCOME MEASURES:

1. Primary Outcome: Enacted Stigma (Intrapersonal)
Description: Change in Enacted Stigma subscore from Substance Use Stigma Mechanisms Scale (SU-SMS) pre- and post-intervention. All responses are given on a 5-point Likert-type scale, with higher scores indicating greater endorsement of substance use stigma. Enacted (6 items) scale can be created by taking the average of the item responses given. Minimum score = 6, Maximum score = 30.
  Reported mean is the change in these scores (pre score - post score), so a positive number for the mean is a reduction in stigma using average scores from the Enacted Stigma subscore.
Time Frame: Immediately before and 2-weeks post-intervention delivery
Population: Intrapersonal arm only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intrapersonal Stigma Reduction
Number analyzed (Participants) | 37
score on a scale | 0.730 (3.813)
Statistical Analysis 1: Comparison: Intrapersonal Stigma Reduction; Pre/post scores within arm; Test type: Other; p = 0.252, t-test, 2 sided

2. Primary Outcome: Anticipated Stigma (Intrapersonal)
Description: Change in Anticipated Stigma subscore from Substance Use Stigma Mechanisms Scale (SU-SMS) pre- and post-intervention. All responses are given on a 5-point Likert-type scale, with higher scores indicating greater endorsement of substance use stigma. Enacted (6 items) scale can be created by taking the average of the item responses given. Minimum score = 6, Maximum score = 30.
  Reported mean is the change in these scores (pre score - post score), so a positive number for the mean is a reduction in stigma using average scores from the Anticipated Stigma subscore.
Time Frame: Immediately before and 2-weeks post-intervention delivery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intrapersonal Stigma Reduction
Number analyzed (Participants) | 37
score on a scale | 0.514 (4.985)
Statistical Analysis 1: Comparison: Intrapersonal Stigma Reduction; Pre/post score within arm; Test type: Other; p = 0.546, t-test, 2 sided

3. Primary Outcome: Internalized Stigma (Intrapersonal)
Description: Change in Internalized Stigma subscore from Substance Use Stigma Mechanisms Scale (SU-SMS) pre- and post-intervention. All responses are given on a 5-point Likert-type scale, with higher scores indicating greater endorsement of substance use stigma. Enacted (6 items) scale can be created by taking the average of the item responses given. Minimum score = 6, Maximum score = 30.
  Reported mean is the change in these scores (pre score - post score), so a positive number for the mean is a reduction in stigma using average scores from the Internalized Stigma subscore.
Time Frame: Immediately before and 2-weeks post-intervention delivery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intrapersonal Stigma Reduction
Number analyzed (Participants) | 37
score on a scale | 2.324 (4.720)
Statistical Analysis 1: Comparison: Intrapersonal Stigma Reduction; Pre/post scores within arm; Test type: Other; p = 0.005, t-test, 2 sided

4. Primary Outcome: Exposure to Drug Users Index Score
Description: Exposure to drug users index includes questions regarding if a participant has been exposed to a drug user at home, at work, at school, etc. (7 items; No = 0, Yes = 1). Score is total count (min score = 0, max score = 7). Higher scores indicate more exposure to drug users.
  Reported mean is the change in this score pre and post intervention (post score - pre score).
Time Frame: Pre/post intervention (week 0)
Population: Interpersonal arm only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interpersonal Stigma Reduction
Number analyzed (Participants) | 21
score on a scale | -0.476 (1.601)
Statistical Analysis 1: Comparison: Interpersonal Stigma Reduction; Pre/post scores within arm; Test type: Other; p = 0.188, t-test, 2 sided

5. Primary Outcome: Drug Use Stigmatization Scale Score
Description: The Drug Use Stigmatization Scale measures stigma against drug users. The scale contains 7 items scored on a 5-point likert scale with higher scores representing higher stigma. The score is the average score of the seven items. Min score = 1, Max score = 5.
  Reported mean is the change in these scores (pre score - post score), so a positive number for the mean is a reduction in stigma.
Time Frame: Pre/post intervention (week 0: post-test immediately followed intervention)
Population: This measure was only given to the Interpersonal arm only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interpersonal Stigma Reduction
Number analyzed (Participants) | 21
score on a scale | 2.105 (4.345)
Statistical Analysis 1: Comparison: Interpersonal Stigma Reduction; Pre/post score within arm; Test type: Other; p = 0.049, t-test, 2 sided

6. Primary Outcome: Stigma of Drug Users Scale Score
Description: The Stigma of Drug Users Scale measures stigma. There are 10 items scored on a 5-point likert scale. Higher scores indicate higher stigma. The score is the average of the 10 items (Min score = 1, Max score = 5).
  The reported mean for this outcome measure is the change in this score pre and post intervention (pre score - post score). A positive mean indicates a reduction in stigma.
Time Frame: Pre/post intervention (week 0: post-test immediately followed intervention)
Population: This measure was only given to the Interpersonal arm only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interpersonal Stigma Reduction
Number analyzed (Participants) | 21
score on a scale | 1.211 (2.323)
Statistical Analysis 1: Comparison: Interpersonal Stigma Reduction; Pre/post scores within arm; Test type: Other; p = 0.036, t-test, 2 sided

7. Secondary Outcome: Engagement in Treatment
Description: Number of participants in intrapersonal arm who made an appointment for treatment after receiving the intervention.
Time Frame: 2-weeks post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intrapersonal Stigma Reduction
Number analyzed (Participants) | 37
Participants | 4

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Intrapersonal Stigma Reduction | Interpersonal Stigma Reduction
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/21
Other Adverse Events (participants affected / at risk) | 0/50 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT04693416/Prot_002.pdf
  • Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/16/NCT04693416/SAP_003.pdf
  • Informed Consent Form (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT04693416/ICF_004.pdf